CLINICAL TRIAL: NCT01670097
Title: A Preliminary Study of Dexamethasone for Dyspnea in Cancer Patients
Brief Title: Dexamethasone Dyspnea Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-0001; NCI-2012-01615 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-01

CONDITIONS: Advanced Cancers; Hematologic Disorder; Solid Tumors
Keywords: Advanced Cancers; Hematologic Disorder; Solid Tumors; Dyspnea; Difficulty breathing; Shortness of breath; Dexamethasone; Decadron; Placebo; Sugar pill; Questionnaires; Surveys; Spirometer; Phone calls
MeSH Terms: conditions — Hematologic Diseases; Dyspnea | interventions — Dexamethasone; Calcium Dobesilate; Sugars; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone 8 mg (2 capsules of 4 mg) given orally twice a day for 4 days, then 4 mg given orally twice a day for 3 days. In the open label phase, patients assigned to either arm asked to take Dexamethasone 4 mg orally twice a day for 7 days. Patient to blow into spirometry machine 1 time a day to test lung function. Questionnaires completed at baseline and at day 7 and 14. It should take about 15 minutes to complete these questionnaires. Questionnaires completed at baseline and at day 7 and 14. It should take about 15 minutes to complete these questionnaires.
  Participants randomized to either dexamethasone or placebo for 7 days in a blinded fashion; this will be followed by an open label phase in which patients in both arms would take dexamethasone for 7 days.
  Interventions: Drug: Dexamethasone; Behavioral: Questionnaires; Device: Spirometer; Other: Phone Calls
- Placebo (Placebo Comparator): Two placebo capsules taken twice a day for 4 days, followed by one capsule twice a day for 3 days. Patient to blow into spirometry machine 1 time a day to test lung function. Questionnaires completed at baseline and at day 7 and 14. It should take about 15 minutes to complete these questionnaires. Questionnaires completed at baseline and at day 7 and 14. It should take about 15 minutes to complete these questionnaires.
  Participants randomized to either dexamethasone or placebo for 7 days in a blinded fashion; this will be followed by an open label phase in which patients in both arms would take dexamethasone for 7 days.
  Interventions: Drug: Dexamethasone; Drug: Placebo; Behavioral: Questionnaires; Device: Spirometer; Other: Phone Calls

INTERVENTIONS:
Drug: Dexamethasone — Group 1 Blinded Phase: 8 mg (2 capsules of 4 mg) given orally twice a day for 4 days, then 4 mg given orally twice a day for 3 days.
  Open Label Phase Groups 1 and 2: 4 mg by mouth twice a day for 7 days.
  Other Names: Decadron
Drug: Placebo — Group 2 Blinded Phase: Two capsules by mouth twice a day for 4 days, followed by one capsule twice a day for 3 days.
  Other Names: Sugar pill
  Arms: Placebo
Behavioral: Questionnaires — Questionnaires completed at baseline and at day 7 and 14. It should take about 15 minutes to complete these questionnaires.
  Other Names: Surveys
Device: Spirometer — Patient to blow into spirometry machine 1 time a day to test lung function.
Other: Phone Calls — Patient called by phone 1 time each day to ask about level of shortness of breath and to remind patient to take capsules. These calls should last about 5 minutes.

SUMMARY:
The goal of this clinical research study is to learn if dexamethasone can help reduce shortness of breath in cancer patients. Researchers also want to learn if it can help to improve lung function and quality of life. In this study, dexamethasone will be compared to a placebo.

Dexamethasone is commonly used for treatment of nausea, tiredness, and pain. It may help patients with shortness of breath.

A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Baseline Tests:

If you are found to be eligible to take part in this study, you will have baseline tests after completing the screening questionnaires. The following tests and procedures will be performed:

* Information will be collected from your medical record about your age, sex, race, disease type, how well you are able to perform the normal activities of daily living, any drugs you are taking, and possible causes of shortness of breath.
* Your breathing rate will be measured.
* The amount of oxygen in your body will be measured using a machine that clips on your finger.
* You will blow into a device called a spirometer a few times to measure your lung function.
* You will be asked to answer 4 questionnaires. The first questionnaire asks you to rate your level of symptoms, such as pain, tiredness, sleep, appetite, depression, anxiety, and drowsiness. The second questionnaire asks about your sensation of breathing. The third questionnaire asks you to rate the intensity of your shortness of breath. The last questionnaire asks about your quality of life. These questionnaires should take a total of about 40 minutes to complete.

Study Groups:

You will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups:

* If you are in Group 1, you will receive dexamethasone.
* If you are in Group 2, you will receive a placebo for 7 days, then dexamethasone for 7 days.

You will have an equal chance of being assigned to either group. Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug/Placebo Administration:

After your baseline tests, you will be given a supply of either the study drug or the placebo to bring home.

Starting the next morning, you will take 2 dexamethasone or placebo capsules twice a day by mouth for 4 days. Then, you will take 1 tablet twice a day for 3 more days.

After the first 7 days, no matter which group you have been assigned to, you will only take 1 dexamethasone capsule twice a day for 7 more days

You should take the capsules around 8 o'clock in the morning and 4 o'clock in the afternoon. You should take the capsules with food and 8 ounces of water.

You will also receive a portable spirometer to test your lung function. You should blow into the machine 1 time a day.

Study Visits/Calls:

On Days 7 and 14, you will return to the clinic or be called by phone. You should bring your capsule boxes with you if you come to the clinic, or have them with you if you are called so the study staff can count the number of capsules. The following tests and procedures will be performed:

* You will be asked to complete the same 4 questionnaires you completed during your baseline tests.
* You will also be asked about any side effects you may be having and if you think the study drug is helping your shortness of breath.
* You will blow into a spirometer to measure your lung function.

During the 14 days you will be taking either the study drug or the placebo on the study, you will be called by phone 1 time each day to ask you about your level of shortness of breath and to remind you to take the capsules. These calls should last about 5 minutes.

Length of Study:

You may continue taking the study drug for up to 14 days, as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if intolerable side effects occur or if you are unable to follow study directions.

Your participation on the study will be over when you have completed the follow-up calls and visit.

This is an investigational study. Dexamethasone is FDA approved and commercially available for the treatment of pain, nausea and tiredness. Its use to help control shortness of breath is investigational.

Up to 40 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer
2. Dyspnea with an average intensity level >3/10 on the numeric rating scale over the past week
3. Clinical or radiologic history of lung/pleural involvement (primary or metastatic), lymphangitic carcinomatosis or airway involvement secondary to tumor infiltration
4. Outpatients at MD Anderson Cancer Center seen by the Supportive Care, Rehabilitation Service, Thoracic Oncology or Pulmonary Medicine
5. Able to communicate in English
6. Karnofsky performance status >=40%
7. Age 18 or older
8. Permission from the attending medical oncologist if the patient is currently on an interventional cancer therapy trial.

Exclusion Criteria:

1. Delirium (i.e. Memorial delirium rating scale >13)
2. Oxygen saturation <90% despite supplemental oxygen >6L/min
3. Previous allergic reactions to dexamethasone
4. Uncontrolled hyperglycemia as defined by any blood glucose of >300 mg/dl in the past two weeks
5. Severe anemia (Hb <7g/L) not corrected prior to study enrollment (bloodwork is not required if patient did not have recent chemotherapy within last 2 weeks)
6. Post-surgical open wound that has not been healed at the time of enrollment
7. Any infection requiring parenteral antibiotics within the past 2 weeks
8. Major surgery within the past 2 weeks
9. Megestrol use at the time of study enrollment
10. Neutropenia (absolute neutrophil count < 1.0) (bloodwork is not required if patient did not have recent chemotherapy within last 2 weeks)
11. Currently on or expected to start cytotoxic chemotherapy with in 1 week of study enrollment
12. Chronic obstructive pulmonary disease (COPD) exacerbation at the time of study enrollment
13. Heart failure exacerbation at the time of study enrollment
14. Chronic systemic corticosteroid use (>14 days) at the time of study enrollment
15. Unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hui D, Kilgore K, Frisbee-Hume S, Park M, Tsao A, Delgado Guay M, Lu C, William W Jr, Pisters K, Eapen G, Fossella F, Amin S, Bruera E. Dexamethasone for Dyspnea in Cancer Patients: A Pilot Double-Blind, Randomized, Controlled Trial. J Pain Symptom Manage. 2016 Jul;52(1):8-16.e1. doi: 10.1016/j.jpainsymman.2015.10.023. Epub 2016 Jun 18. PMID 27330023
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult cancer patient with lung involvement were recruited between 1/2013 and 5/2015 from the Supportive Care Center outpatient clinic of MD Anderson Cancer Center who satisfied the inclusion and exclusion criteria.
Pre-assignment Details: A total of 52 participants enrolled for this study. Among them, 41 patients were randomized. 6 participants declined to continue and 5 participants became ineligible (3 started steroids, 2 had other reasons) before randomization, thus a total of 11 participants were dropped out before randomization.
Groups:
- Intervention Group (Dexamethasone): Received Dexamethasone capsule 8 mg twice daily for 4 days, then 4 mg capsule twice daily for 3 days. It was followed by dexamethasone capsule 4 mg twice daily for 7 days.
- Controlled Group (Placebo): Received Placebo for 7 days, It was followed by dexamethasone capsule 4 mg twice daily for 7 days.
Period: Overall Study
Arm/Group | Intervention Group (Dexamethasone) | Controlled Group (Placebo)
Started | 20 | 21
Completed Week 1 Intervention | 18 | 17
Completed Week 2 Intervention | 13 | 15
Completed | 18 | 17
Not Completed | 2 | 4
Not completed — Started Phase 1 cancer treatment | 1 | 0
Not completed — Study burden | 1 | 0
Not completed — COPD exacerbation | 0 | 1
Not completed — Neutropenia | 0 | 1
Not completed — Clinical deterioration | 0 | 1
Not completed — Disease progression | 0 | 1

BASELINE CHARACTERISTICS:
Population: Data included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Dexamethasone) | Controlled Group (Placebo) | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Median (Full Range); unit: years] | 62 [49 to 71] | 64 [48 to 78] | 63 [48 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41
Education [Count of Participants; unit: Participants]
  High School or less | 16 | 18 | 34
  College and above | 4 | 3 | 7
Cancer Type [Count of Participants; unit: Participants]
  Mesothelioma | 1 | 3 | 4
  Non-small cell lung cancer | 14 | 17 | 31
  Small cell lung cancer | 2 | 0 | 2
  Other | 3 | 1 | 4
Cancer Stage [Count of Participants; unit: Participants]
  Localized | 4 | 1 | 5
  Locally advanced | 3 | 4 | 7
  Metastatic/recurrent | 13 | 16 | 29
Comorbidities [Count of Participants; unit: Participants]
  COPD | 2 | 7 | 9
  Asthma | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed the Dyspnea Numeric Rating Scale
Description: Number of participants who completed the dyspnea numeric rating scale on Day 7
Time Frame: Baseline to Day 7
Population: Baseline Analysis included all randomized participants, 20 participants in intervention arm and 21 participants in control arm
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (Dexamethasone) | Controlled Group (Placebo)
Number analyzed (Participants) | 20 | 21
Participants | 18 | 17

2. Secondary Outcome: Edmonton Symptom Assessment System Dyspnea Score
Description: The Secondary outcome is the Edmonton Symptom Assessment System dyspnea intensity which is measured with a single 11-point numeric rating score that ranges between 0 and 10, with 0 being no symptom at all and 10 being worst possible. We measured the change in Edmonton Symptom Assessment System dyspnea numeric rating score (average 24 h) form baseline to Day 4, Day 7 and Day 14.
Time Frame: Baseline to Day 4, Day 7, Day 14
Population: The number of participants varied by milestone study days (Baseline (38 participants) , Day 4 (30 participants) , Day 7 (30 participants) and Day 14 (28 participants) who completed the Edmonton Symptom Assessment Questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group (Dexamethasone) | Controlled Group (Placebo)
Number analyzed (Participants) | 19 | 19
score on a scale
  Day 4: number analyzed (Participants) | 15 | 15
  Day 4 | -1.9 [-3.3 to -0.5] | -0.7 [-2.1 to 0.6]
  Day 7: number analyzed (Participants) | 16 | 14
  Day 7 | -1.8 [-3.2 to -0.3] | -1.3 [-2.4 to -0.2]
  Day 14: number analyzed (Participants) | 13 | 15
  Day 14 | -2.1 [-3.5 to -0.6] | -1.7 [-2.7 to -0.7]

3. Secondary Outcome: Dyspnea Numeric Rating Score (Now)
Description: Secondary outcome was dyspnea intensity 'now' using a dyspnea numeric rating scale that ranges from 0 (no shortness of breath) to 10 (worst possible shortness of breath). We measured the change in Dyspnea numeric rating score form baseline to Day 4, Day 7 and Day 14.
Time Frame: Baseline to day 4, Day 7 and Day 14
Population: The number of participants varied by milestone study days (Baseline (38 participants), Day 4, (35 participants) Day 7 (35 participants), and Day 14 (26 participants) who completed the Dyspnea Numeric Rating Score Questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group (Dexamethasone) | Controlled Group (Placebo)
Number analyzed (Participants) | 19 | 19
score on a scale
  Day 4: number analyzed (Participants) | 18 | 17
  Day 4 | 0 [-1 to 1] | -0.1 [-1.1 to 1]
  Day 7: number analyzed (Participants) | 18 | 17
  Day 7 | -1.1 [-2.4 to 0.2] | -0.2 [-1.6 to 1.2]
  Day 14: number analyzed (Participants) | 12 | 14
  Day 14 | -1.6 [-3 to -0.2] | -1.5 [-2.5 to -0.5]

4. Secondary Outcome: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core- 30 Dyspnea
Description: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30, consists of 30 items that encompasses three symptom scales (pain, fatigue, nausea/vomiting), six single-item symptom items, five functional scales (physical, cognitive, role, emotional, and social), and one scale assessing global health status/quality of life. Each scale comprises 2-5 items. All items have four response categories (1=not at all, 2=a little, 3=quite a bit, 4=very much), except for two items assessing overall health status/quality of life, which use a seven-point scale. This questionnaire includes one item to assess dyspnea during the past week ("Were you short of breath?). The four-point ordinal scale was transformed to 0-100 points using a formula, higher scores indicate worse dyspnea. We measured the change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core- 30 Dyspnea score form baseline to Day 4, Day 7 and Day 14.
Time Frame: Baseline to day 4, Day 7 and Day 14.
Population: The number of participants varied by milestone study days (Baseline (38 participants), Day 4 (30 participants), Day 7 (29 participants), and Day 14 (28 participants) who completed the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-20 Dyspnea.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group (Dexamethasone) | Controlled Group (Placebo)
Number analyzed (Participants) | 19 | 19
score on a scale
  Day 4: number analyzed (Participants) | 15 | 15
  Day 4 | -15.6 [-29.3 to -1.8] | 0 [-14 to 14]
  Day 7: number analyzed (Participants) | 16 | 13
  Day 7 | -10.4 [-21.1 to 0.3] | -5.1 [-19 to 8.8]
  Day 14: number analyzed (Participants) | 13 | 15
  Day 14 | -7.7 [-22.3 to 6.9] | -6.7 [-19.2 to 5.8]

ADVERSE EVENTS:
Time Frame: Baseline to Day 4, Day 7, and Day 14.
Description: As open label medication (Dexamethasone capsules 4 mg twice daily for 7 days) was given to both 'Intervention group' and 'Controlled group' after the initial study medication, we did not measure or looked for the adverse events for open label medication (the last 7 days). We measured the adverse events only for the first 7 days when the intervention and controlled group received 2 different study medications.
Groups:
- Intervention Group (Dexamethasone): Received Dexamethasone capsule 8 mg twice daily for 4 days, then 4 mg capsule daily for 3 days. It was followed by dexamethasone capsule 4 mg twice daily for 7 days.
Arm/Group | Intervention Group (Dexamethasone) | Controlled Group (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 3/20 | 5/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Group (Dexamethasone) (N=20) | Controlled Group (Placebo) (N=21)
Anxiety/Irritability (Nervous system disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Halitosis (Gastrointestinal disorders) | 1 | 0
Edema (General disorders) | 3 | 1
Hiccup (Nervous system disorders) | 1 | 0
Hot flash (Nervous system disorders) | 1 | 0
Hyperglycemia (Gastrointestinal disorders) | 1 | 1
Hyperhidrosis (Nervous system disorders) | 1 | 0
Insomnia (General disorders) | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Blurred vision (Nervous system disorders) | 0 | 2
Fatigue (General disorders) | 0 | 3
Flasing (Nervous system disorders) | 0 | 1
Mouth sores (Gastrointestinal disorders) | 0 | 1
Taste changes (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Nausea/vomiting (Gastrointestinal disorders) | 0 | 4
Pain (Nervous system disorders) | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastric Hemorrhage (Gastrointestinal disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT01670097/Prot_SAP_000.pdf